CLINICAL TRIAL: NCT01047111
Title: A Phase Ⅲ Study of Left Side Thoracotomy Approach (Sweet Procedure) Versus Right Side Thoracotomy Plus Midline Laparotomy Approach (Ivor-Lewis Procedure) Esophagectomy in Middle or Lower Third Intrathoracic Esophageal Cancer
Brief Title: Esophagectomy: Sweet Versus Ivor-Lewis (ESVIL) (ECTOP-2001)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fudan University (Other)
Responsible Party: Principal Investigator, Haiquan Chen, Chief, Department of thoracic surgery, Fudan University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 201001ECFD
Record Dates: First submitted 2010-01-11; First posted 2010-01-12 (Estimated); Last update posted 2023-07-20 (Actual); Status verified 2023-07

CONDITIONS: Esophageal Neoplasms
Keywords: Esophageal Neoplasms; Esophagectomy
MeSH Terms: conditions — Esophageal Neoplasms | interventions — Esophagectomy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Ivor-Lewis Procedure (Active Comparator): Arm A: Esophagectomy was conducted through right side thoracotomy plus midline laparotomy approach:Ivor-Lewis Procedure.
  Interventions: Procedure: Esophagectomy
- Sweet Procedure (Active Comparator): Arm B: Esophagectomy was conducted through left side thoracotomy or thoracoabdominal incision: Sweet Procedure
  Interventions: Procedure: Esophagectomy

INTERVENTIONS:
Procedure: Esophagectomy — Esophagectomy Through Right Side Thoracotomy plus Midline Laparotomy Approach: Ivor-Lewis Procedure VS Esophagectomy Through Left Side Thoracotomy Approach: Sweet Procedure
  Other Names: Right side approach esophagectomy; Left side approach esophagectomy

SUMMARY:
This is a clinical trial from Eastern Cooperative Thoracic Oncology Project (ECTOP), numbered as ECTOP-2001. Esophageal carcinoma is an aggressive disease with a poor prognosis. Surgical resection remains the basic method of management of this malignancy. Although different approaches have been described for the surgical resection of esophageal cancer, there is no statistical evidence based on large scale prospective randomized trials with regard to the issue that which is the optimal surgical approach for esophageal cancer. The purpose of this study is to test two different approach of transthoracic esophagectomy (Right Side Thoracotomy plus Midline Laparotomy Approach: Ivor-Lewis Procedure and Left Side Thoracotomy Approach: Sweet Procedure) in middle or lower third intrathoracic esophageal cancer. This research is being done to see whether one approach is superior than the other approach with better long-term outcome and acceptable postoperative short-term outcome or not.

DETAILED DESCRIPTION:
Background :

Esophageal carcinoma is an aggressive disease with a poor prognosis. Surgical resection remains the basic method of management of this malignancy. Although different approaches have been described for the surgical resection of esophageal cancer, there is no statistical evidence based on large scale prospective randomized trials with regard to the issue that which is the optimal surgical approach for esophageal cancer. In middle or lower third intrathoracic esophageal cancer, a great number of thoracic surgeon preferred the Ivor-Lewis Procedure(Right Side Thoracotomy plus Midline Laparotomy Approach), and believe that this approach can get better exposure for the upper mediastinal node dissection so can get the better long-term survival. But some others preferred the Sweet Procedure(Left Side Thoracotomy Approach),especially in china, more than two of the third unit performed the left side approach esophagectomy routinely and the long-term survival was reported equal to even better than the right side approach. The purpose of this study is to conduct a large scale prospective randomized Phase Ⅲ clinical trial to test that based on the long-term outcomes(overall survival and disease free survival )and postoperative short-term outcomes(mortality, morbidity),whether one approach is superior than the other approach or not.

Objectives:

1. To compare overall survival after right side approach and left side approach esophagectomy
2. To compare locoregional recurrence, disease free survival after right side approach and left side approach esophagectomy
3. To compare postoperative morbidity and mortality in the two groups
4. To evaluate short and long term quality of life after the two procedures

Design: Prospective randomized controlled

Setting: Fudan University Cancer Center, Shanghai, China.

Patients and methods : All patients with biopsy proven carcinoma of the middle or lower third of the esophagus presenting to our hospital will be considered for the study.

Staging investigations will be standard and will include

1. Computed Tomography (CT) scans in all patients
2. Esophagogastroscopy
3. Barium swallow
4. Endoscopic Ultrasonography (EUS) wherever possible
5. PET-CT scan wherever possible

Randomization:

Block randomization will be done using a computer generated sheet. Randomization will be performed 3 days to 1 week before the operation.

All surgeries will be performed under general anesthesia with epidural analgesia. The surgery will be either performed by or under the direct supervision of consultant thoracic surgeons with experience in esophageal surgery. Operative time, blood loss, blood product replacement and all intraoperative details will be recorded in the proforma. Patients will be shifted postoperatively to the intensive care unit (ICU) for observation and subsequently to the recovery or high dependency ward once stabilized. Postoperative details including period of postoperative ventilation, hemorrhage, pulmonary and cardiac complications, arrhythmias, thoracic duct leak, anastomotic leak, wound infection and recurrent laryngeal nerve paresis or palsy will be recorded. Postoperative mortality will be defined as 30-day mortality plus death before discharge after surgery. The total duration of ICU stay and hospital stay will also be recorded.

Follow up:

Patients will be followed up three monthly for the first two years and six monthly for the third to fifth years and annually thereafter. A detailed history and clinical examination and CT scan, barium swallow and ultrasound will be done routinely on every follow up.

Data management: All collected data will be entered into a statistical software package for subsequent analysis

Main research variables:

Primary end point: Disease free survival in the two arms

Secondary endpoints:

1. Overall survival
2. Locoregional recurrence
3. Postoperative morbidity and mortality
4. Quality of life : assessed with EORTC QLQ-C30 scale and EORTC QLQ- OES18 scale.

ELIGIBILITY:
Inclusion Criteria:

* Patients with histologically proven squamous cell esophageal cancer
* Patients with cT1-T3/N0-N1 mid or distal third (inferior to carina and 3cm superior to cardia ) operable esophageal lesion. Staging investigations including esophagogastroscopy, chest and abdominal CT scan, barium swallow and selective endoscopic ultrasonography showing no evidence of invading adjacent structure such as spine, bronchus, pericardium , descending aorta and without enlargement cervical and celiac nodes (diameter of short axis greater than 1.5cm) measured at CT scans.
* Karnofsky performance status greater than or equal to 80%
* Pulmonary and cardiac function must be acceptable for surgery according to institutional standards.
* Acceptable hepatic, renal and bone marrow function

Exclusion Criteria:

* Patients with low performance status(Karnofsky score <80%)
* Past history of malignancy
* Stage investigations indicating unresectable advanced disease(T4 or M1a,M1b)
* Patients with any other serious underlying medical condition that would impair the ability of the patient to receive or comply with protocol treatment
* Patients medically unfit for surgical resection
* Patients with pulmonary reserve inadequate to undergo thoracotomy and extensive mediastinal lymphadenectomy.
* Patients with a significant history of unstable cardiovascular disease that in the opinion of the treating physician should preclude the patient from protocol treatment.
* Uncontrolled diabetes mellitus or uncontrolled infection, including HIV or interstitial pneumonia or interstitial fibrosis.
* Significant psychiatric illness that would interfere with patient compliance
* Patients with severe hepatic cirrhosis or with serious renal disease unacceptable for surgery
* Patients considered of salvage surgery after definitive chemoradiotherapy
* Patients after neoadjuvant chemoradiotherapy
* Patients above the age of 75 years
* Patients unreliable for follow up

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Actual)
Dates: Start 2010-05; Primary Completion 2012-07 (Actual); Study Completion 2017-07 (Actual)

PRIMARY OUTCOMES:
Disease free survival | 6 years

SECONDARY OUTCOMES:
Overall survival | 6 years
postoperative morbidity and mortality | 3 years
Locoreginal recurrence and recurrence pattern | 6 years

CONTACTS AND LOCATIONS:
Overall Officials: Haiquan Chen, MD, Principal Investigator — Fudan University
Locations (1):
- Fudan University Cancer Center, Shanghai, Shanghai Municipality, China

REFERENCES:
- [Derived] Li B, Xiang J, Zhang Y, Li H, Zhang J, Sun Y, Hu H, Miao L, Ma L, Luo X, Chen S, Ye T, Zhang Y, Zhang Y, Chen H. Comparison of Ivor-Lewis vs Sweet esophagectomy for esophageal squamous cell carcinoma: a randomized clinical trial. JAMA Surg. 2015 Apr;150(4):292-8. doi: 10.1001/jamasurg.2014.2877. PMID 25650816